CLINICAL TRIAL: NCT02964247
Title: LIRA-ADD2SGLT2i - Liraglutide Versus Placebo as add-on to SGLT2 Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-4315; U1111-1184-8086 (Other: WHO)
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- liraglutide + SGLT2i ± metformin (Experimental)
  Interventions: Drug: liraglutide
- liraglutide placebo + SGLT2i ± metformin (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Liraglutide given s.c. once daily, gradually titrated to 1.8 mg/day as an add-on to the subject's stable pre-trial SGLT2 inhibitor ± metformin for 26 weeks
  Arms: liraglutide + SGLT2i ± metformin
Drug: placebo — Liraglutide placebo given s.c. once daily, gradually titrated to 1.8 mg/day as an add-on to the subject's stable pre-trial SGLT2 inhibitor ± metformin for 26 weeks
  Arms: liraglutide placebo + SGLT2i ± metformin

SUMMARY:
The trial is conducted in Asia, Europe, North America and South America. The aim of the study is to compare the effect of liraglutide 1.8 mg/day versus placebo as add-on to an SGLT2 inhibitor with or without metformin on glycaemic control in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male or female, age 18 years or older at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus.
* HbA1c of 7.0-9.5% (53-80 mmol/mol) (both inclusive).
* Stable dose of an SGLT-2 inhibitor as monotherapy or in combination (including fixed-dose drug combination) with a stable dose of metformin (1500 mg or more, or maximum tolerated dose) for at least 90 days prior to the day of screening. All medications in compliance with current local label.
* Body mass index of 20 kg/m^2 or above.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice).
* History of diabetic ketoacidosis while being treated with SGLT2 inhibitors.
* Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of less than 60 mL/min/1.73m^2 as defined by Kidney Disease Improving Global Outcomes (KDIGO) classification using isotope dilution mass spectrometry (IDMS) for serum creatinine measured at screening.
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 90 days prior to the day of screening. However, short term insulin treatment for a maximum of 14 days during the 90 days prior to screening is allowed.
* Family or personal history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma. Family is defined as a first degree relative.
* History or presence of pancreatitis (acute or chronic).
* Impaired liver function, defined as ALT 2.5 or more times upper normal limit at screening.
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (50):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Montgomery, Alabama
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Vista, California
  - Novo Nordisk Investigational Site, Gainesville, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Maitland, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Miami Lakes, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Statesboro, Georgia
  - Novo Nordisk Investigational Site, Blackfoot, Idaho
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Rochester, Michigan
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Kinston, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, McMurray, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Moncks Corner, South Carolina
  - Novo Nordisk Investigational Site, Mt. Pleasant, South Carolina
  - Novo Nordisk Investigational Site, Myrtle Beach, South Carolina
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Edinburg, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Humble, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Schertz, Texas
  - Novo Nordisk Investigational Site, Spokane, Washington
- Brazil (3):
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, Porto Alegre, Rio Grande do Sul
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
- India (9):
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Coimbatore, Tamil Nadu
  - Novo Nordisk Investigational Site, Hyderabad, Telangana
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi
- Israel (4):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Novo Nordisk Investigational Site, Ponce, Puerto Rico
- Novo Nordisk Investigational Site, Saint Petersburg, Russia
- United Arab Emirates (3):
  - Novo Nordisk Investigational Site, Al Ain City
  - Novo Nordisk Investigational Site, Dubai
  - Novo Nordisk Investigational Site, Umm Al Quwain City

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Blonde L, Belousova L, Fainberg U, Garcia-Hernandez PA, Jain SM, Kaltoft MS, Mosenzon O, Nafach J, Palle MS, Rea R. Liraglutide as add-on to sodium-glucose co-transporter-2 inhibitors in patients with inadequately controlled type 2 diabetes: LIRA-ADD2SGLT2i, a 26-week, randomized, double-blind, placebo-controlled trial. Diabetes Obes Metab. 2020 Jun;22(6):929-937. doi: 10.1111/dom.13978. Epub 2020 Feb 14. PMID 31984646
- [Derived] Blonde L, Fainberg U, Kaltoft MS, Mosenzon O, Ramesh C, Rea R. Efficacy of liraglutide added to sodium-glucose cotransporter-2 inhibitors in type 2 diabetes, stratified by baseline characteristics: Post-hoc analysis of LIRA-ADD2SGLT2i. Diabetes Obes Metab. 2021 Oct;23(10):2234-2241. doi: 10.1111/dom.14464. Epub 2021 Jul 8. PMID 34132018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 74 sites in 7 countries. All the sites have screened and randomised subjects. Brazil: 3 sites, India: 7 sites, Israel: 6 sites, Mexico: 2 sites, Russian Federation: 3 sites, United Arab Emirates: 5 sites, United States: 48 sites screened and randomised subjects.
Groups:
- Liraglutide: Eligible subjects were given liraglutide subcutaneously (s.c.), once daily (OD) for 26 weeks. Subjects received 0.6 mg dose of liraglutide in week 1, dose was escalated to 1.2 mg in week 2 and 1.8 mg in week 3. Subjects remained on the stable dose of 1.8 mg liraglutide from week 3 to 26. Subjects continued their pre-trial SGLT2 inhibitor as monotherapy or in combination with metformin at stable pre-trial dose. Any one of three SGLT2 inhibitors were allowed as pre-trial therapy: Invokana®, Farxiga®/Forxiga® and Jardiance®. Stable pre-trial treatment with metformin was defined as ≥1500 mg/day or at the maximum tolerated dose. Any fixed dose combination of SGLT2 inhibitors and metformin was also allowed in this trial as background medication.
  A follow-up visit was scheduled one week after the end of treatment.
- Placebo: Eligible subjects were given liraglutide placebo subcutaneously (s.c.), once daily (OD) for 26 weeks. Dose escalation for placebo matched that for liraglutide with regards to volume. Subjects remained on the stable dose of 1.8 mg placebo from week 3 to 26. Subjects continued their pre-trial SGLT2 inhibitor as monotherapy or in combination with metformin at stable pre-trial dose during the trial. Any one of three SGLT2 inhibitors were allowed as pre-trial therapy: Invokana®, Farxiga®/Forxiga® and Jardiance®. Stable pre-trial treatment with metformin was defined as ≥1500 mg/day or at the maximum tolerated dose. Any fixed dose combination of SGLT2 inhibitors and metformin was also allowed in this trial as background medication.
  A follow-up visit was scheduled one week after the end of treatment.
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 203 | 100
Exposed to Trial Product | 202 | 100
Completed | 200 | 98
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) includes all randomised subjects. Subjects in the FAS contribute to the evaluation 'as randomised'.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Placebo | Total
Number analyzed (Participants) | 203 | 100 | 303
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.72 (10.08) | 56.03 (9.89) | 55.15 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 42 | 120
  Male | 125 | 58 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 35 | 94
  Not Hispanic or Latino | 144 | 65 | 209
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 38 | 15 | 53
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 5 | 17
  White | 131 | 59 | 190
  Other | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change from baseline (week 0) to week 26 in glycosylated haemoglobin was evaluated for 2 different observation period 'in-trial' observation period and 'on-treatment without rescue medication" observation period. The 'in-trial' observation period represents the time-period where subjects were considered to be in the trial, regardless of whether or not the subjects had initiated rescue medication or prematurely discontinued trial product. The 'on-treatment' observation period is the part of the in-trial observation period during which subjects were treated with the trial product, that is the time from the first dose to the last dose of trial product. The 'on-treatment without rescue medication' observation period is a part of 'on-treatment' observation period during which subjects were considered treated with trial product and had not initiated any rescue medications.
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
Percentage of HbA1c
  in-trial obs. period: number analyzed (Participants) | 195 | 95
  in-trial obs. period | -1.00 (0.86) | -0.32 (0.83)
  on-treatment without rescue medication obs. period: number analyzed (Participants) | 179 | 80
  on-treatment without rescue medication obs. period | -1.05 (0.85) | -0.35 (0.80)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Statistical analysis for the primary estimand. Primary estimand: treatment effect (effectiveness) based on the FAS using week 26 measurements from the in-trial observation period. The change in HbA1c from baseline to week 26 were analysed using a pattern mixture model with multiple imputation to impute missing data, with treatment, country and the stratification factor (metformin use at baseline: yes vs. no) as categorical fixed effects and baseline HbA1c as covariate; Test type: Superiority; p < .001, pattern mixture model; Treatment difference = -0.68, 95% CI 2-sided [-0.89 to -0.48], Standard Error of Mean 0.10 — Liraglutide - Placebo
Statistical Analysis 2: Comparison: Liraglutide vs Placebo; Statistical analysis for the secondary estimand.The change in HbA1c from baseline up to and including week 26 at scheduled time points were analysed using MMRM with treatment, country and the stratification factor (metformin use at baseline: yes vs. no) as categorical fixed effects and baseline HbA1c as covariate, all nested within visit; Test type: Superiority — Test was not controlled for type I error. Secondary estimand: treatment effect (efficacy) based on the FAS using post baseline measurements up to and including week 26 from the on-treatment without rescue medication obs. period; p < .001, Mixed Models Analysis; Treatment difference = -0.74, 95% CI 2-sided [-0.94 to -0.53], Standard Error of Mean 0.10 — Liraglutide - Placebo

2. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) to week 26 in body weight was evaluated for 2 different observation period 'in-trial' observation period and 'on-treatment without rescue medication" observation period. The 'in-trial' observation period represents the time-period where subjects were considered to be in the trial, regardless of whether or not the subjects had initiated rescue medication or prematurely discontinued trial product. The 'on-treatment' observation period is the part of the in-trial observation period during which subjects were treated with the trial product, that is the time from the first dose to the last dose of trial product. The 'on-treatment without rescue medication' observation period is a part of 'on-treatment' observation period during which subjects were considered treated with trial product and had not initiated any rescue medications.
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
Kg
  in-trial obs. period: number analyzed (Participants) | 196 | 97
  in-trial obs. period | -2.84 (3.83) | -2.02 (3.32)
  on-treatment without rescue medication obs. period: number analyzed (Participants) | 182 | 82
  on-treatment without rescue medication obs. period | -2.89 (3.81) | -2.09 (2.96)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Statistical analysis for the primary estimand. Primary estimand: treatment effect (effectiveness) based on the FAS using week 26 measurements from the in-trial observation period. The change in body weight from baseline to week 26 were analysed using a pattern mixture model with multiple imputation to impute missing data, with treatment, country and the stratification factor (metformin use at baseline: yes vs. no) as categorical fixed effects and baseline body weight as covariate; Test type: Superiority; p = 0.077, pattern mixture model; Treatment difference = -0.82, 95% CI 2-sided [-1.73 to 0.09], Standard Error of Mean 0.46 — Liraglutide - Placebo
Statistical Analysis 2: Comparison: Liraglutide vs Placebo; Statistical analysis for the secondary estimand. The change in body weight from baseline up to and including week 26 at scheduled time points were analysed using MMRM with treatment, country and the stratification factor (metformin use at baseline: yes vs. no) as categorical fixed effects and baseline body weight as covariate, all nested within visit; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.062, Mixed Models Analysis; Treatment difference = -0.86, 95% CI 2-sided [-1.77 to 0.04], Standard Error of Mean 0.46 — Liraglutide - Placebo

3. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change from baseline (week 0) to week 26 in fasting plasma glucose ('in-trial' observation period)
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Mean (Standard Deviation); unit: milligram/dL
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
milligram/dL | -27.00 (35.01) | -11.97 (45.20)

4. Secondary Outcome: Subjects Who Achieve HbA1c Below 7.0% (53 mmol/Mol), American Diabetes Association Target
Description: Percentage of subjects who achieve HbA1c below 7.0% (53 mmol/mol), American Diabetes Association target, after 26 weeks ('in-trial' observation period)
Time Frame: Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 195 | 95
Percentage of Participants
  Yes | 51.79 | 23.16
  No | 48.21 | 76.84

5. Secondary Outcome: Subjects Who Achieve HbA1c Below or Equal to 6.5% (48 mmol/Mol), American Association of Clinical Endocrinologists Target
Description: Percentage of subjects who achieve HbA1c below or equal to 6.5% (48 mmol/mol), American Association of Clinical Endocrinologists target, after 26 weeks ('in-trial' observation period)
Time Frame: Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 195 | 95
Percentage of Participants
  Yes | 34.36 | 9.47
  No | 65.64 | 90.53

6. Secondary Outcome: Subjects Who Achieve HbA1c Below 7.0% (53 mmol/Mol) Without Severe or Blood Glucose Confirmed Symptomatic Hypoglycaemia Episodes and no Weight Gain.
Description: Percentage of subjects who achieve HbA1c below 7.0% (53 mmol/mol) without severe or blood glucose confirmed symptomatic hypoglycaemia episodes and no weight gain, after 26 weeks ('in-trial' observation period)
Time Frame: Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 195 | 94
Percentage of Participants
  Yes | 47.69 | 19.15
  No | 52.31 | 80.85

7. Secondary Outcome: Subjects Who Achieve HbA1c Reduction Above or Equal to 1% (11mmol/Mol) and Weight Loss Above or Equal to 3%.
Description: Percentage of subjects who achieve HbA1c reduction above or equal to 1% (11mmol/mol) and weight loss above or equal to 3%, after 26 weeks ('in-trial' observation period)
Time Frame: Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 195 | 94
Percentage of Participants
  Yes | 29.74 | 7.45
  No | 70.26 | 92.55

8. Secondary Outcome: Change in Self-measured Plasma Glucose 7-point Profile - Mean 7-point Profile
Description: Change in self-measured plasma glucose 7-point profile - mean 7-point profile after 26 weeks. Subjects were instructed to measure their plasma glucose at following 7 timepoints: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, at bedtime. Mean of the 7-point profile was calculated ('in-trial' observation period).
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Mean (Standard Deviation); unit: milligram/dL
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
milligram/dL | -33.93 (37.17) | -18.85 (40.81)

9. Secondary Outcome: Change in Self-measured Plasma Glucose 7-point Profile - Mean Post Prandial Increments (Over All Meals)
Description: Subjects were instructed to measure their plasma glucose at following 7 timepoints: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, at bedtime. The mean increment over all meals was derived as the mean of all available meal increments ('in-trial' observation period)
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Mean (Standard Deviation); unit: milligram/dL
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
milligram/dL | -11.06 (41.29) | -4.44 (44.77)

10. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Observed mean change from baseline (week 0) to week 26 in body mass index (BMI). BMI was calculated based on body weight and height ('in-trial' observation period)
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
kg/m^2 | -1.02 (1.40) | -0.72 (1.20)

11. Secondary Outcome: Subjects Who Achieve HbA1c Below 7.0% (53 mmol/Mol) and no Weight Gain
Description: Percentage of subjects who achieve HbA1c below 7.0% (53 mmol/mol) and no weight gain, after 26 week ('in-trial' observation period).
Time Frame: Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 195 | 94
Percentage of Participants
  Yes | 47.69 | 19.15
  No | 52.31 | 80.85

12. Secondary Outcome: Subjects Who Achieve HbA1c Below 7.0% (53 mmol/Mol), no Weight Gain and Systolic Blood Pressure Below 140 mmHg.
Description: Percentage of subjects who achieve HbA1c below 7.0% (53 mmol/mol), no weight gain and systolic blood pressure below 140 mmHg, after 26 weeks ('in-trial' observation period)
Time Frame: Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 195 | 94
Percentage of Participants
  Yes | 42.05 | 18.09
  No | 57.95 | 81.91

13. Secondary Outcome: Subjects Who Achieve HbA1c Reduction Above or Equal to 1% (11mmol/Mol)
Description: Percentage of subjects who achieve HbA1c reduction above or equal to 1% (11mmol/mol), after 26 weeks ('in-trial' observation period)
Time Frame: Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 195 | 95
Percentage of Participants
  Yes | 52.31 | 16.84
  No | 47.69 | 83.16

14. Secondary Outcome: Subjects Who Achieve HbA1c Reduction Above or Equal to 1% (11mmol/Mol) and no Weight Gain
Description: Percentage of subjects who achieve HbA1c reduction above or equal to 1% (11mmol/mol) and no weight gain, after 26 weeks.
Time Frame: Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 195 | 94
Percentage of Participants
  Yes | 45.13 | 14.89
  No | 54.87 | 85.11

15. Secondary Outcome: Number of Treatment Emergent Adverse Events
Description: The on-treatment summary of adverse events includes treatment-emergent events with onset on or after the first day of exposure to randomised treatment and no later than the minimum of the date of the follow-up visit or the last day of randomised treatment + 7 days or the date of last subject-investigator contact.
Time Frame: Week 0 - 26 + 7 days
Population: Safety analysis set (SAS) includes all subjects exposed to at least one dose of trial product. Subjects in the SAS contribute to the evaluation based on the trial product received for the period they were on-treatment, referred to as contributing to the evaluation 'as treated'. 'Number Analyzed' = subjects with available data.
Measure: Number; unit: Events
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 202 | 100
Events | 426 | 106

16. Secondary Outcome: Number of Treatment Emergent Severe or Blood Glucose Confirmed Symptomatic Hypoglycaemia Episodes
Description: Treatment emergent hypoglycaemic episode is defined episode with onset on or after the first day of exposure to randomised treatment and no later than the minimum of the date of the follow-up visit or the last day of randomised treatment + 1 days or the date of last subject-investigator contact. Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to American Diabetes Association's (ADA) classification or blood glucose confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Severe hypoglycaemia according to the ADA definition: an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions.
Time Frame: Week 0 - 26
Population: as for outcome 15
Measure: Number; unit: Episodes
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 202 | 100
Episodes | 0 | 3

17. Secondary Outcome: Change in Fasting Blood Lipids - Total Cholesterol
Description: Fasting total cholesterol measured in mg/dL. Observed mean change in fasting total cholesterol from baseline (week 0) to week 26 is presented as ratio to baseline value.
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
Ratio | 0.95 (45.1) | 0.99 (42.3)

18. Secondary Outcome: Change in Fasting Blood Lipids - Low Density Lipoprotein (LDL) Cholesterol
Description: Low density lipoprotein (LDL) cholesterol measured in mg/dL. Observed mean change in fasting low density lipoprotein cholesterol from baseline (week 0) to week 26 is presented as ratio to baseline value.
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
Ratio | 0.97 (58.6) | 1.01 (54.1)

19. Secondary Outcome: Change in Fasting Blood Lipids - High Density Lipoprotein (HDL) Cholesterol
Description: High density lipoprotein (HDL) cholesterol measured in mg/dL. Observed mean change in fasting high density lipoprotein cholesterol from baseline (week 0) to week 26 is presented as ratio to baseline value.
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
Ratio | 1.05 (41.4) | 1.01 (39.7)

20. Secondary Outcome: Change in Fasting Blood Lipids - Very Low Density Lipoprotein (VLDL) Cholesterol
Description: Very low density lipoprotein (VLDL) cholesterol measured in mg/dL. Observed mean change in fasting very low density lipoprotein cholesterol from baseline (week 0) to week 26 is presented as ratio to baseline value.
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
Ratio | 0.83 (69.0) | 0.94 (64.5)

21. Secondary Outcome: Change in Fasting Blood Lipids-triglycerides
Description: Fasting triglycerides measured in mg/dL. Observed mean change in fasting triglycerides from baseline (week 0) to week 26 is presented as ratio to baseline value.
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
Ratio | 0.81 (71.5) | 0.93 (70.0)

22. Secondary Outcome: Change in Fasting Blood Lipids- Free Fatty Acids (FFA)
Description: Free fatty acids measured in mg/dL. Observed mean change in fasting free fatty acids from baseline (week 0) to week 26 is presented as ratio to baseline value.
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
Ratio | 0.80 (86.6) | 0.86 (92.0)

23. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) to week 26 in waist circumference ('in-trial' observation period).
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
cm | -4.28 (11.19) | -1.77 (4.42)

24. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change from baseline (week 0) in systolic blood pressure after 26 weeks ('in-trial' observation period).
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
mmHg | -1.95 (13.42) | -3.35 (12.36)

25. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change from baseline (week 0) in diastolic blood pressure after 26 weeks ('in-trial' observation period).
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 203 | 100
mmHg | -0.72 (8.04) | -1.12 (8.55)

26. Secondary Outcome: Subjects Who Achieve Weight Loss by 3% or More
Description: as for outcome 7
Time Frame: Week 26
Population: Full analysis set (FAS) includes all randomised subjects. 'Number Analyzed' = subjects with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 196 | 97
Percentage of participants
  Yes | 46.43 | 41.24
  No | 53.57 | 58.76

ADVERSE EVENTS:
Time Frame: Week 0 (randomisation visit) to week 26 (end-of-treatment visit) + 7 days
Description: Treatment emergent adverse event is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product. Safety analysis set includes all subjects exposed to at least one dose of trial product.
Arm/Group | Liraglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/202 | 0/100
Serious Adverse Events (participants affected / at risk) | 5/202 | 1/100
Other Adverse Events (participants affected / at risk) | 87/202 | 8/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=202) | Placebo (N=100)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Eyelid cyst (Eye disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=202) | Placebo (N=100)
Constipation (Gastrointestinal disorders) | 18 (19) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 19 (19) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 19 (24) | 3 (3)
Nausea (Gastrointestinal disorders) | 53 (61) | 6 (8)
Vomiting (Gastrointestinal disorders) | 17 (20) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT02964247/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT02964247/SAP_001.pdf